CLINICAL TRIAL: NCT03118375
Title: Hearing Outcomes Using Super-power Processors in Bone Anchored Implant Recipients
Brief Title: Super Power in BAI
Status: Terminated | Type: Observational
Why Stopped: Could not adequately recruit enough subjects to reach appropriate sample size
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Hillary A Snapp, Assistant Professor, University of Miami
Other Study IDs: 20170083
Record Dates: First submitted 2017-04-12; First posted 2017-04-18 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Conductive and Sensorineural Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Cohort: Hearing and speech tests will be performed on the subject and repeated to compare results obtained using their current BAHA processor against results using super-power BAHA processor.
  Interventions: Device: super-power BAHA processor

INTERVENTIONS:
Device: super-power BAHA processor — The super-power BAHA processor will be provided for use at the study visit only to run different types of hearing tests, speech understanding tests in quiet, and speech understanding tests in noise. The same tests will be performed with the use of the subject's current BAHA processor for comparison.

SUMMARY:
The purpose of this study is to assess the benefit of new super-power bone-anchored hearing aid (BAHA) processors in BAHA users. BAHAs are able to help people with mixed/conductive and single-sided hearing loss when they are unable to use or receive limited benefit from traditional hearing. Until recently, BAHAs were only recommended to people with up to a moderate hearing loss. New super-power BAHA processors may be able to help people who previously were not candidates for BAHAs or received limited benefit from them. The information collected in this study may lead to improved evaluation of and expanded treatment options for people considering BAHA. Different types of hearing tests will be used to compare the devices.

DETAILED DESCRIPTION:
The objective of this study is to assess the benefit of new super-power bone-anchored hearing aid (BAHA) processors in BAHA users. BAHAs are able to help people with mixed/conductive and single-sided hearing loss when they were not receiving benefit from traditional hearing aids or could not use them due to differences in their ears related to surgery or congenital anomalies. Stronger super-power processors may be able to help individuals who previously did not meet candidacy for BAHA. This study will evaluate how much benefit they are getting from their current devices compared to new super-power devices.

The information collected in this study may lead to improved evaluation of patients considering BAHA implantation and expanded treatment options for new and existing BAHA users. Primary outcome measures will include hearing threshold and speech perception measures. All devices are commercially available and FDA approved.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* meet candidacy criteria for a high gain super-power processor with a fitting range up to 65 dB
* native English speaker

Exclusion Criteria:

* do not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult bone-anchored implant recipients who met candidacy criteria for a high gain super-power processor with a fitting range up to 65 dB.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2017-04-29 (Actual); Study Completion 2017-04-29 (Actual)

PRIMARY OUTCOMES:
Threshold testing | 1 hour
  Conventional hearing test will be performed. Sound field testing will be performed to establish aided thresholds using the individual's current BAHA processor and super power BAHA processor
Speech perception in noise | 1 hour
  Speech perception in noise will be evaluated without hearing devices and then using the individual's current BAHA processor and super power BAHA processor
Speech perception in quiet | 1 hour
  Word understanding will be evaluated without hearing devices and then using the individual's current BAHA processor and super power BAHA processor

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Snapp, AuD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Department of Otolaryngology, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arehart KH, Kates JM, Anderson MC, Harvey LO Jr. Effects of noise and distortion on speech quality judgments in normal-hearing and hearing-impaired listeners. J Acoust Soc Am. 2007 Aug;122(2):1150-64. doi: 10.1121/1.2754061. PMID 17672661
- [Background] Flynn MC, Sadeghi A, Halvarsson G. Baha solutions for patients with severe mixed hearing loss. Cochlear Implants Int. 2009;10 Suppl 1:43-7. doi: 10.1179/cim.2009.10.Supplement-1.43. PMID 19195004
- [Background] Gantz BJ, Turner C, Gfeller KE, Lowder MW. Preservation of hearing in cochlear implant surgery: advantages of combined electrical and acoustical speech processing. Laryngoscope. 2005 May;115(5):796-802. doi: 10.1097/01.MLG.0000157695.07536.D2. PMID 15867642
- [Background] Yu JK, Wong LL, Tsang WS, Tong MC. A tutorial on implantable hearing amplification options for adults with unilateral microtia and atresia. Biomed Res Int. 2014;2014:703256. doi: 10.1155/2014/703256. Epub 2014 Jun 2. PMID 24991564
- [Background] Norman, J. (2015). Review of fitting ranges. Cochlear Bone Anchored Solutions AB. D773528
- [Background] Rubinstein JT, Parkinson WS, Tyler RS, Gantz BJ. Residual speech recognition and cochlear implant performance: effects of implantation criteria. Am J Otol. 1999 Jul;20(4):445-52. PMID 10431885
- [Background] Verhaegen VJ, Mulder JJ, Mylanus EA, Cremers CW, Snik AF. Profound mixed hearing loss: bone-anchored hearing aid system or cochlear implant? Ann Otol Rhinol Laryngol. 2009 Oct;118(10):693-7. doi: 10.1177/000348940911801002. PMID 19894395